CLINICAL TRIAL: NCT05225935
Title: Computed Tomography-Guided Catheter Ablation for Ventricular Tachycardia (InEurHeart Study)
Brief Title: Computed Tomography-Guided Catheter Ablation for Ventricular Tachycardia
Acronym: InEurHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: EIT Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2021/61
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Ventricular Tachycardia
Keywords: Myocardial infarction; Ventricular Tachycardia; Catheter Ablation; Imaging; Cardiac computed tomography
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- image-guided VT ablation strategy (Experimental): Catheter ablation procedure performed as part of standard care, although with the addition of an image-based 3D heart model including detailed anatomy and primary ablation targets
  Interventions: Device: image-guided VT ablation strategy
- conventional VT ablation strategy (Active Comparator): Catheter ablation performed using conventional mapping techniques to identify targets. The ablation strategy will be left to the local investigator's decision, based on the clinical scenario and operator's habits.
  Interventions: Device: conventional VT ablation strategy

INTERVENTIONS:
Device: image-guided VT ablation strategy — Catheter ablation procedure performed as part of standard care, although with the addition of an image-based 3D heart model including detailed anatomy and primary ablation targets
  Arms: image-guided VT ablation strategy
Device: conventional VT ablation strategy — Catheter ablation will be performed using conventional mapping techniques to identify targets. The ablation strategy will be left to the local investigator's decision, based on the clinical scenario and operator's habits.
  Arms: conventional VT ablation strategy

SUMMARY:
This double arm randomized study will compare 2 ventricular tachycardia ablation strategies: the standard strategy based on invasive substrate and VT mapping with 3D electro-anatomical system vs a tailored strategy which identifies targets based on pre-procedural CT-scan imaging. The primary endpoint will be procedure duration and secondary endpoints will include safety and efficacy criteria as well as medico-economic evaluation.

DETAILED DESCRIPTION:
Ventricular tachycardia ablation is a non-drug alternative for patients with recurrent VT and ischemic cardiomyopathy with a class 1 indication in the latest guidelines. However, it is poorly standardised and reserved to expert centres. Proof of concept studies have demonstrated that image-guided VT ablation is feasible, and that it may improve the efficiency of VT ablation.

Ablation strategy no longer relying on intracardiac 2-dimensional surface catheter measurements for target identification, but on 3- dimensional pre-operative images of the myocardium acquired by computed tomography (CT) would shorten the procedure, make it more reproducible and less dependent of the operator's experience without altering efficacy.

This randomized study will compare VT ablation based on substrate/VT isthmus identification via intracardiac catheter vs identification via pre-procedural CT-scan. Ablation will be performed with the same material.

Primary endpoint will be procedure duration. Secondary endpoints will compare efficacy and safety of both strategies as well as cost-effectiveness.

Expected results are a reduction procedure duration, without alteration of the efficacy for the CT-guided procedure with an improved medico-economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Indication for catheter ablation intervention with planned preoperative cardiac CT scan
* Prior myocardial infarction (using the international definition of MI: Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non- ischemic cause with documentation of prior ischemic injury),
* Presence of an implantable cardioverter defibrillator, or planned ID implantation before discharge, and
* One of the following monomorphic VT events within last 6 months:

  * A: ≥3 episodes of VT treated with antitachycardia pacing (ATP),
  * B: ≥1 appropriate ICD shocks,
  * C: sustained VT below detection rate of the ICD documented by ECG or any cardiac monitor
  * D: Sustained VT recorded on 12 leads ECG in the absence of ICD
* Highly effective contraception for women of childbearing potential, maintained during research procedures
* Signed informed consent ,
* Affiliated to or beneficiary of a health insurance

Exclusion Criteria:

* Unable to understand the nature, risks, significance and implications of the clinical investigation or unwilling to provide written informed consent,
* Active ischemia (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of VT (e.g. drug-induced arrhythmia), had recent acute coronary syndrome within 30 days thought to be due to acute coronary arterial thrombosis, or have CCS functional class IV angina. Note that biomarker level elevation alone after ventricular arrhythmias does not denote acute coronary syndrome or active ischemia,
* Are known to have protruding left ventricular thrombus or mechanical aortic and mitral valves,
* Have had a prior catheter ablation procedure for VT,
* Presenting arrhythmia: polymorphic VT or ventricular fibrillation (VF),
* Renal failure (Creatinine clearance <30 mL/min), have NYHA Functional class IV heart failure, or a systemic illness likely to limit survival to <1 year,
* Women who are pregnant, lactating, or who are planning to become pregnant during the anticipated study period,
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Procedure duration | Day 1
  Procedure duration measured from the first introduction of a catheter in the cardiac chamber of interest (mainly left ventricle or epicardial space) to the end of the last radiofrequency application

SECONDARY OUTCOMES:
Number of VT | Baseline, Month 6, , Month 12
  Number of VT
Appropriate antitachycardia pacing from ICD >14 days after procedure | Month 1, Month 6, Month 12
  Number of appropriate antitachycardia pacing from ICD >14 days after procedure. for ventricular arrhythmia
Appropriate ICD shock >14 days after procedure | Month 1, Month 6, Month 12
  Number of any appropriate ICD shock >14 days after procedure. The ICD shocks will be automatically recorded through the device logs and transmitted via remote monitoring whenever possible. Appropriate ICD therapies are defined as antitachycardia pacing or shock delivered
Inappropriate ICD shock >14 days after procedure | Month 1, Month 6, Month 12
  Number of any inappropriate ICD shock >14 days after procedure. The ICD shocks will be automatically recorded through the device logs and transmitted via remote monitoring whenever possible. - Inappropriate ICD therapies are defined as antitachycardia pacing or shock delivered for anything but ventricular arrhythmia
Electrical storm >14 days after procedure | Month 1, Month 6, Month 12
  Number of electrical storm >14 days after procedure. Electrical storm is defined as 3 episodes of sustained VT/VF within 24 hours
Sustained VT not treated by ICD >14 days after procedure | Month 1, Month 6, Month 12
  Number of sustained VT not treated by ICD >14 days after procedure
anti-arrhythmic drugs | Month 1, Month 6, Month 12
  Use of anti-arrhythmic drugs >30 days after procedure
Death | Month 12
  Death
General health-related quality of life | Baseline, Month 1, Month 6, Month 12
  Quality of life using EQ-5D-5L questionnaire: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Additinonally, the questionnaire records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Radiofrequency (RF) applications | Day 1
  Proportion of Radiofrequency (RF) applications within isthmii identified by CT-Scan vs outside isthmii
Societal healthcare costs | Month 1, Month 3, Month 6, Month 9, Month 12
  Total one-year healthcare costs from a societal perspective : Cumulative over 12 months with medical consumption, informal care, and absence from work, all measured according to the time frame indicated down below
Payer healthcare costs | Month 1, Month 3, Month 6, Month 9, Month 12
  Total one-year healthcare costs from a payer's perspective: Cumulative over 12 months with medical consumption, measured according to the time frame indicated down below
Quality-adjusted life | Month 1, Month 3, Month 6, Month 9, Month 12
  Number of (quality-adjusted life-QALY) years: Cumulative over 12 months with EQ-5D-5L measured according to the time frame indicated down below
Incremental cost per QALY gained | Month 1, Month 3, Month 6, Month 9, Month 12
  Incremental cost per QALY gained (ratio): 12-month cumulative costs divided by 12-month cumulative QALYs
Incremental cost per VT episode avoided | Month 1, Month 3, Month 6, Month 9, Month 12
  Incremental cost per VT episode avoided (ratio): 12-month cumulative costs divided by cumulative number of VT in 12-months
Incremental cost per additional day without a VT episode | Month 1, Month 3, Month 6, Month 9, Month 12
  Incremental cost per additional day without a VT episode (ratio): 12-month cumulative costs divided by cumulative number of days without VT in 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Sacher, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (14):
- Austria (2):
  - Medical University of Graz, Graz
  - Public Hospital Elisabethinen Linz, Linz
- France (5):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Limoges, Limoges
  - APHP Salpétrière, Paris
  - CHU de Bordeaux, Pessac
  - CHU de Toulouse, Toulouse
- Germany (5):
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Rhön-Klinikum AG, Bad Neustadt an der Saale
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Deutsches Herzzentrum München, München
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - Vaudois University Hospital, Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided